CLINICAL TRIAL: NCT01633879
Title: Health and Success: Addressing Proven Factors in HIV Prevention for Latino Youth
Brief Title: Addressing Proven Factors in HIV Prevention for Latino Youth
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Education Development Center, Inc. (Industry)
Responsible Party: Principal Investigator, Lydia O'Donnell, Senior Scientist, Education Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD062084 (NIH)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: HIV; Sexually Transmitted Infections
Keywords: parenting, prevention, HIV/AIDS, adolescents, Latino
MeSH Terms: conditions — Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome | interventions — Health; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- parent education (Experimental): audio-CD parent EDC supporting positive parenting practices
  Interventions: Behavioral: audio-CD parent education
- parent and school intervention (Experimental): health and success parent and school intervention
  Interventions: Behavioral: health and success parent and school
- print materials (No Intervention): brochures to parents

INTERVENTIONS:
Behavioral: audio-CD parent education — audio CD stories in English and Spanish that support positive parenting practices
  Other Names: health and success
  Arms: parent education
Behavioral: health and success parent and school — Parenting education and school intervention
  Arms: parent and school intervention

SUMMARY:
This study tests the effectiveness of the bilingual Health and Success program, which aims to support Latino parents and schools in their efforts to promote the academic success and healthy choices of youth, with the goal of reducing barriers that lead to elevated levels of HIV/AIDS in urban Latino communities.

ELIGIBILITY:
Inclusion Criteria:

* youth attend school selected as study site
* youth in 6-7th grade

Exclusion Criteria:

* parent/youth non-English or Spanish speakers

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3400 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
reduction in risk behavior | 18 months
  The study will examine whether there is a reduction in risky sexual behavior among youth exposed to the two treatment conditions compared to the control condition.